CLINICAL TRIAL: NCT04735042
Title: Use of Combination Empagliflozin/Linagliptin or Dapagliflozin/Saxagliptin vs Empagliflozin or Dapagliflozin Alone, Subclinical Inflammation of the Genito-urinary Tract and Risk of Infections.
Brief Title: SGLT-2 and DPP-4 Inhibition, Subclinical Inflammation of the Genito-urinary Tract and Risk of Infections.
Acronym: UTI-flog
Status: Completed | Type: Observational
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Anna Solini, Associate Professor, University of Pisa
Other Study IDs: AS0005
Record Dates: First submitted 2021-01-22; First posted 2021-02-02 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Type 2 Diabetes; Urinary Tract Infections
Keywords: UTI; Type 2 Diabetes; SGLT2 inhibitors; DPP4 inhibitors
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Urinary Tract Infections | interventions — empagliflozin; Linagliptin; dapagliflozin; saxagliptin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum Urine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- SGLT2 and DPP-4 inhibitors: Patients undergoing SGLT2i and DPP4i.
  Interventions: Drug: Empagliflozin / Linagliptin or Dapagliflozin/Saxagliptin Pill
- SGLT2 inhibitors only: Patients undergoing SGLT2i alone.
  Interventions: Drug: Empagliflozin or Dapagliflozin Pill

INTERVENTIONS:
Drug: Empagliflozin / Linagliptin or Dapagliflozin/Saxagliptin Pill — association between SGLT2-inhibitor and DPP4-inhibitor
  Other Names: Glyxambi or Qtern
  Groups: SGLT2 and DPP-4 inhibitors
Drug: Empagliflozin or Dapagliflozin Pill — SGLT2-inhibitor: diabetic oral drug with diuretic properties.
  Other Names: Jardiance or Forxiga
  Groups: SGLT2 inhibitors only

SUMMARY:
In this observational study, 60 subjects with type 2 diabetes (T2D) and eligible, as per good clinical practice, for therapy with SGLT-2 inhibitor, will be randomized to receive a SGLT-2 inhibitor or a fixed dose combination of SGLT-2 inhibitor with a DPP4-inihibitor for 12 weeks. Measures will be performed at baseline and after 12 weeks of treatment, as per good clinical practice.

DETAILED DESCRIPTION:
The day of the study patients undergo a routine clinical evaluation. Whole blood samples will be collected from an antecubital vein to assess serum/plasma aliquots of 200 μl each (frozen at -80°C until required for quantitation) for evaluation of biochemical parameters (fasting glucose, HbA1c, lipid profile, serum creatinine, uric acid, electrolytes, liver function enzymes, albumin).

A mid-stream first urine in the morning sample will be collected into a sterile container. 50 ml of urine will be immediately transferred into a sterile falcon and centrifugated at 4500 rpm for 10 min. After removal of the supernatant and addition of 10 ml of PBS or sterile physiological solution, the sample will be further centrifugated at 4500 rpm for 10 min. The supernatant will be removed and the pellet stored in a falcon at -80°C.

Genomic DNA will be extracted throw Qiamp DNA mini kit (QIAGEN) and quantified using spectrophotometric assay.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes diagnosis
* Hb1Ac ≥ 7% and ≤ 9%

Exclusion Criteria:

* Hb1Ac > 9%
* current treatment with an SGLT2i or a DPP4i drugs, or in the prior 4 week
* irritating and/or obstructive urinary or genital symptoms
* menstrual cycle for women
* current antibiotic treatment or in the prior 4 weeks
* anatomical or functional abnormalities of the urinary tract (e.g. incontinence, neurological bladder, bladder prolapse).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will consecutively enrolled 60 patients among those referring to the Departiment of Diabetes and Metabolic disease, Santa Chiara Hospital, Pisa.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-10-07 (Actual); Primary Completion 2021-10-07 (Actual); Study Completion 2022-04-07 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in metagenomic analysis based on rRNA 16S gene | Each patients will be analyzed at baseline and after 12 weeks
  Metagenomic analysis based on rRNA 16S gene will be performed by Novogene on Illumina platform (Hong Kong, China)
Change from Baseline of total bacterial load | Each patients will be analyzed at baseline and after 12 weeks
  Absolute quantification of total bacterial load in the original sample using real-Time quantitative PCR

SECONDARY OUTCOMES:
Fasting glucose | baseline and 12 week
  Fasting glucose measured in a fasting morning blood sample
Glycated Haemoglobin | baseline and 12 week
  HbA1c in a fasting measured in a morning blood sample
Renal function | baseline and 12 week
  Using creatinine measured in a fasting morning blood sample and estimated by eGFR (calculated with the CDK-EPI formula)
Albumin excretion | baseline and 12 week
  Measured by urinary albumin/creatinine ratio
Total cholesterol | baseline and 12 week
  Total cholesterol measured in a fasting morning blood sample
HDL cholesterol | baseline and 12 week
  HDL cholesterol measured in a fasting morning blood sample
Triglycerides | baseline and 12 week
  Triglycerides measured in a fasting morning blood sample

CONTACTS AND LOCATIONS:
Overall Officials: Anna Solini, MD, PhD, Principal Investigator — University of Pisa
Locations (1):
- University of Pisa, Pisa, Pisa, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nitzan O, Elias M, Chazan B, Saliba W. Urinary tract infections in patients with type 2 diabetes mellitus: review of prevalence, diagnosis, and management. Diabetes Metab Syndr Obes. 2015 Feb 26;8:129-36. doi: 10.2147/DMSO.S51792. eCollection 2015. PMID 25759592
- [Background] Renko M, Tapanainen P, Tossavainen P, Pokka T, Uhari M. Meta-analysis of the significance of asymptomatic bacteriuria in diabetes. Diabetes Care. 2011 Jan;34(1):230-5. doi: 10.2337/dc10-0421. Epub 2010 Oct 11. PMID 20937688
- [Background] Schmiemann G, Kniehl E, Gebhardt K, Matejczyk MM, Hummers-Pradier E. The diagnosis of urinary tract infection: a systematic review. Dtsch Arztebl Int. 2010 May;107(21):361-7. doi: 10.3238/arztebl.2010.0361. Epub 2010 May 28. PMID 20539810
- [Background] He K, Hu Y, Shi JC, Zhu YQ, Mao XM. Prevalence, risk factors and microorganisms of urinary tract infections in patients with type 2 diabetes mellitus: a retrospective study in China. Ther Clin Risk Manag. 2018 Feb 26;14:403-408. doi: 10.2147/TCRM.S147078. eCollection 2018. PMID 29520146
- [Background] Aswani SM, Chandrashekar U, Shivashankara K, Pruthvi B. Clinical profile of urinary tract infections in diabetics and non-diabetics. Australas Med J. 2014 Jan 31;7(1):29-34. doi: 10.4066/AMJ.2014.1906. eCollection 2014. PMID 24567764
- [Background] Masajtis-Zagajewska A, Nowicki M. New markers of urinary tract infection. Clin Chim Acta. 2017 Aug;471:286-291. doi: 10.1016/j.cca.2017.06.003. Epub 2017 Jun 13. PMID 28622967
- [Background] Liu J, Li L, Li S, Jia P, Deng K, Chen W, Sun X. Effects of SGLT2 inhibitors on UTIs and genital infections in type 2 diabetes mellitus: a systematic review and meta-analysis. Sci Rep. 2017 Jun 6;7(1):2824. doi: 10.1038/s41598-017-02733-w. PMID 28588220
- [Background] Li D, Wang T, Shen S, Fang Z, Dong Y, Tang H. Urinary tract and genital infections in patients with type 2 diabetes treated with sodium-glucose co-transporter 2 inhibitors: A meta-analysis of randomized controlled trials. Diabetes Obes Metab. 2017 Mar;19(3):348-355. doi: 10.1111/dom.12825. Epub 2016 Dec 19. PMID 27862830
- [Background] Yu H, Woo VC. Emerging use of combination therapies for the management of type 2 diabetes - focus on saxagliptin and dapagliflozin. Diabetes Metab Syndr Obes. 2017 Jul 21;10:317-332. doi: 10.2147/DMSO.S117982. eCollection 2017. PMID 28769579
- [Background] Del Prato S, Rosenstock J, Garcia-Sanchez R, Iqbal N, Hansen L, Johnsson E, Chen H, Mathieu C. Safety and tolerability of dapagliflozin, saxagliptin and metformin in combination: Post-hoc analysis of concomitant add-on versus sequential add-on to metformin and of triple versus dual therapy with metformin. Diabetes Obes Metab. 2018 Jun;20(6):1542-1546. doi: 10.1111/dom.13258. Epub 2018 Mar 25. PMID 29446523
- [Background] Kim NH, Yu T, Lee DH. The nonglycemic actions of dipeptidyl peptidase-4 inhibitors. Biomed Res Int. 2014;2014:368703. doi: 10.1155/2014/368703. Epub 2014 Jul 21. PMID 25140306
- [Background] Lewis DA, Brown R, Williams J, White P, Jacobson SK, Marchesi JR, Drake MJ. The human urinary microbiome; bacterial DNA in voided urine of asymptomatic adults. Front Cell Infect Microbiol. 2013 Aug 15;3:41. doi: 10.3389/fcimb.2013.00041. eCollection 2013. PMID 23967406